CLINICAL TRIAL: NCT01202474
Title: A Study of Effectiveness and Safety of Apidra in Combination With Lantus Therapy in Basal-bolus Insulin Regimen in Inadequately Controlled Children and Adolescents With Type 1 Diabetes in the Russian Federation.
Brief Title: Apidra Children & Adolescents Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_04884; U1111-1116-8645 (Other: UTN)
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Glargine

ARMS (1):
- insulin glulisine and insulin glargine (Experimental): insulin glulisine and insulin glargine basal/bolus regimen in accordance with the summary of product characteristics and titrated to Plasma glucose target as defined by American Diabetes Association (ADA) recommendations age-specific goals (12)
  Interventions: Drug: INSULIN GLULISINE; Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLULISINE — Pharmaceutical form: solution for injection Route of administration: subcutaneous Dose regimen: once a day
  Other Names: Apidra
Drug: INSULIN GLARGINE — Pharmaceutical form:solution for injection Route of administration: subcutaneous Dose regimen: 0-15 minutes before meal or within 20 minutes from the start of meal according to prandial plasma glucose values
  Other Names: Lantus

SUMMARY:
Primary Objective:

Evaluate the percentage of patients achieving glycosylated hemoglobin (HbA1c) level < 8% (in patients of 6-12 years old) and HbA1c level < 7.5% (in patients of 13-17 year old) at 6 and 12 months of treatment

Secondary Objectives:

Change in HbA1c level at 6 and 12 months of treatment Monthly rate of hypoglycaemia/per patient from the baseline to the end of the study Change in daily dose of glargine and glulisine at 6 and 12 months of treatment.

ELIGIBILITY:
Inclusion criteria:

* ChildrenAdolescents with Type 1 diabetes Mellitus l(T1DM) onger than 1 year duration
* Age 6 -17 y.o.
* With 8%<HbA1c <10%
* Treated with insulin glargine and any rapid insulin
* Ability to perform a self blood-glucose monitoring (SBGM)
* Signed Informed consent.

Exclusion criteria:

* Diabetes Mellitus type 2
* ChildrenAdolescents with Type 1 diabetes Mellitus previously treated with Apidra
* Hypersensitivity to Insulin glulisine
* Pregnant or lactation women
* Gestational diabetes mellitus
* Treatment with systemic corticosteroids in the 1 month prior to study entry
* T1DM complications: such as already existing active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before study entry or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving HbA1c level < 8% (in patients 6-12 year-old) and HbA1c level < 7.5 % (in patients 13-17 year-old) | at 6 and 12 months of treatment

SECONDARY OUTCOMES:
Change in HbA1c plasma level | at 6 and 12 months of treatment
Monthly rate of hypoglycaemia | from baseline to 12 months of treatment (study cut off)
Change in daily dose of glargine and glulisine | at 6 and 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative office, Moscow, Russia